CLINICAL TRIAL: NCT00004827
Title: Study of Docosahexaenoic Acid (DHA) Supplementation in Patients With X-Linked Retinitis Pigmentosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13351; RFS-FDR001232
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-05

CONDITIONS: Retinitis Pigmentosa
Keywords: ophthalmologic disorders; rare disease; retinitis pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa; Rare Diseases | interventions — Docosahexaenoic Acids

INTERVENTIONS:
Drug: docosahexaenoic acid

SUMMARY:
OBJECTIVES:

I. Evaluate the potential of nutritional docosahexaenoic acid (DHA) supplementation to normalize the level of DHA in red blood cells, and to retard the progression of visual function loss in patients with early stage X-linked retinitis pigmentosa.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, parallel, double blind study. Patients receive 2 gel capsules per day of either docosahexaenoic acid (DHA) enriched oil or a placebo oil. Oral DHA supplementation continues daily for 3 years.

All patients are followed every 6 months for the 3 year duration of the study.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of X-linked retinitis pigmentosa

Early stage disease Sufficient cone function determined by recordable ERG (30 Hz amplitude; greater than 0.32 microvolts) Visual fields greater than 20 degrees Sufficient rod function (greater than 3.0 microvolts amplitude)

Media clarity sufficient for fundus photography

--Prior/Concurrent Therapy--

No concurrent use of anticoagulant medication

--Patient Characteristics--

* No chronic metabolic disease that may interfere with fatty acid metabolism
* No bleeding of clinical significance

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46
Dates: Start 1996-03; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Dennis R. Hoffman, Study Chair — Retina Foundation of the Southwest

REFERENCES:
- [Derived] Schwartz SG, Wang X, Chavis P, Kuriyan AE, Abariga SA. Vitamin A and fish oils for preventing the progression of retinitis pigmentosa. Cochrane Database Syst Rev. 2020 Jun 18;6(6):CD008428. doi: 10.1002/14651858.CD008428.pub3. PMID 32573764